CLINICAL TRIAL: NCT04119167
Title: Use of Growth Differentiation Factor 15 as a Biomarker for Early Diagnosis of Diabetes Mellitus and Monitoring of Progress of Diabetic Peripheral Neuropathy in Asians
Brief Title: Use of GDF15 as a Biomarker for Early Diagnosis of DM and Monitoring of Progress of Complications in Asians
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201900948B0
Record Dates: First submitted 2019-09-22; First posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Polyneuropathy; Diabetic Nephropathies
Keywords: Diabetes Mellitus, Type 2; Diabetic Polyneuropathy; Diabetic Nephropathy; Growth Differentiation Factor 15
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Neuropathies; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Significant differences in the expression of individual Growth Differentiation Factor 15 (GDF-15) proteins among Taiwanese harboring different mitochondrial genotypes are noted, and their blood serum levels also exhibited associations with diabetes. GDF-15 was originally discovered as an autocrine regulator of macrophage activation and shown to play important roles in fibrosis, malignancy, cardiovascular disease, glycemic control, and obesity. However, the relationship between GDF-15 and pre-diabetes and diabetes in Asian populations has yet to be fully investigated. Besides, any indirect associations between GDF-15 levels and diabetic complications remain unclear. The investigators aim to further investigate the role of GDF-15 levels in the initial diagnosis of diabetes, the monitoring of medication effectiveness and disease progression, and related complications such as diabetic nephropathy and neuropathy. The DNA isolated from the blood samples will be evaluated to determine individual mitochondria haplogroups, including variants located within the coding and control regions of the mitochondrial genome.

DETAILED DESCRIPTION:
Previous studies have confirmed that mitochondria are associated with insulin resistance or diabetes. As the prevalence of type 2 diabetes mellitus (T2DM) continues to increase worldwide, early detection and intervention of diabetes can extend life expectancy, reduce complications and decrease medical expenses.

Significant differences in the expression of individual Growth Differentiation Factor 15 (GDF-15) proteins among Taiwanese harboring different mitochondrial genotypes are noted, and their blood serum levels also exhibited associations with diabetes. However, the relationship between GDF-15 and pre-diabetes and diabetes in Asian populations has yet to be fully investigated. In addition, any indirect associations between GDF-15 levels and diabetic complications remain unclear.

The investigators propose a two-year study project to elucidate several hot topics, including the level of GDF-15 in the initial diagnosis of diabetes in Asians if the interpretation is affected by drugs, and whether it is related to the progression of diabetes and related complications, such as diabetic nephropathy or peripheral neuropathy. By investigating mitochondrial genomic variations and the expression of related proteins, The investigators can determine the significant level of GDF-15 in the initial diagnosis of diabetes, medication effects, and diabetic complications. The DNA isolated from the blood samples will be evaluated by Luminex or Sanger sequencing method to determine individual mitochondria haplogroups, including variants located within the coding and control regions of the mitochondrial genome. The investigators aim to establish the significance of GDF-15 testing in Asian hyperglycemic populations. Our research is expected to have a positive impact on improving the early detection and interventional effectiveness of diabetes treatments, thereby reducing the financial burden on the global healthcare system.

The investigators plan to recruit patients, including 250 participants with pre-DM or DM and 250 participants as the control group. The investigators will enroll patients >20 years old and pregnant women will be excluded. Moving from the above considerations, the investigators will collect clinical information and lifestyle habits (smoking, alcohol consumption, physical activity, etc.) prospectively and review the medical records of these patients, who has newly-diagnosed impaired fasting glucose (IFG) or DM at the Chang Gung Memorial Hospital- Kaohsiung Medical Center since May, 2019. It takes about 1 year to collect the patient's specimen and data gradually, and the experiment takes about 1 year. For volunteers participating in the study, there is only a risk in the blood draw process.

For privacy protection and confidentiality, the investigators set a research code representing each participant's identity. This code will not display the name, identification number, and address. For the results and medical records, the Principal Investigator will carefully maintain privacy. If any research result is published, the participant's identity will remain confidential.

GDF15 is a non-glucose protein, and only one fasting blood sample is needed. Serum GDF15 level is stable at room temperature for 48 hours, with consistent value despite four freeze/thaw cycles (20 hours at -70°C followed by 4 hours at room temperature). The anticoagulant used for sampling does not affect the measurements. One factor affecting the interpretation of GDF15 is pregnancy. In a study about the association between GDF15 and pregnancy and hyperemesis gravidarum, the association between the genes GDF15 and IGFBP7 and hyperemesis was found. GDF15 is highly expressed in placental trophoblast cells and its protein appears to promote placentation via activation of neurons in the hypothalamus and area postrema (vomiting center) of the brainstem. IGFBP7 also plays a role in placentation, appetite, and cachexia. Therefore, circulating the GDF15 level is affected by the state of pregnancy. That's why the investigators will exclude pregnant women in our study.

After the research team explains the protocol and review of the informed consent form (The Institutional Review Board No. 201900948B0C601, informed consent form Version 3). The patient has all the questions answered and signed consent prior to any study procedure. A copy of the signed consent will be given to the patient. The samples of blood count and the extracted DNA will be measured within one year, including the haplogroup, the mitochondrial gene single set, and mitochondrial control region and binding gene variant. The storage location is the tissue bank of Kaohsiung Medical Center of Chang Gung Memorial Hospital.

ELIGIBILITY:
Inclusion Criteria:

* adult participants with age >20, with pre-DM or DM as the study group and participants without hyperglycemia as the control group

Exclusion Criteria:

* Pregnant woman or who is under breastfeeding
* Who is difficult to understand or sign the informed consent
* With coagulopathy or hematologic disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From the outpatient department of internal medicine at the Chang Gung Memorial Hospital- Kaohsiung Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Level of GDF15 | Up to 9 months
  Level of serum GDF15 (pg/mL)
Complication of diabetes | Up to 9 months
  Neuropathy (the finding of Nerve Conduction Velocity), retinopathy (the finding of non-mydriatic fundoscopy), nephropathy (the level of serum Creatinine and the amount of albuminuria), number of Participants with coronary artery disease, cerebrovascular disease
Level of glycated hemoglobin (HbA1c) | Up to 9 months
  glycemic control (%)
Level of fasting blood sugar | Up to 9 months
  glycemic control (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Wen Weng, MD/PhD, Principal Investigator — Assistant Professor of Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Currently in the submission stage, and we will then share with other researchers after publication.